CLINICAL TRIAL: NCT03320980
Title: Split-in-situ Resection With Radio-frequency Ablation Instead of Liver Partition on the First Stage (RALPPS) in Patients With Hilar and Intrahepatic Cholangiocarcinoma
Brief Title: RALPPS in Patients With Hilar and Intrahepatic Cholangiocarcinoma
Status: Completed | Type: Observational
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Other Study IDs: MCNC 09/2017
Record Dates: First submitted 2017-10-10; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hilar Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma
Keywords: ALPPS; RALPPS; Portal Vein Embolization; Hilar Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RALPPS: Patients with initial volume of FLR < 40% which underwent RALPPS and major liver resection (as the second stage of RALPPS) for hilar and intrahepatic cholangiocarcinoma
  Interventions: Procedure: RALPPS
- Portal vein embolization (PVE): Patients with initial volume of FLR < 40% undergoing PVE and major liver resection for hilar and intrahepatic cholangiocarcinoma
  Interventions: Procedure: portal vein embolization + major liver resection

INTERVENTIONS:
Procedure: RALPPS — RALPPS: split-in-situ resection with radio-frequency ablation (RFA) instead of liver partition on the first stage and major liver resection on the second stage
  Groups: RALPPS
Procedure: portal vein embolization + major liver resection — PVE on the first stage and major liver resection on the second stage
  Groups: Portal vein embolization (PVE)

SUMMARY:
Unsatisfactory immediate outcomes of Associating liver partition and portal vein ligation for staged hepatectomy (ALPPS) in surgery of cholangiocarcinoma suggested that patients with biliary cancer should not be treated by ALPPS. Short-term results of ALPPS variants with reduced surgical trauma on the first stage in patients with cholangiocarcinoma were not yet estimated. The objective of the study was estimation of the short-term results of split-in-situ resection with radio-frequency ablation (RFA) instead of liver partition on the first stage (RALPPS) in patients with hilar (h-CCA) and intrahepatic (i-CCA) cholangiocarcinoma compared with portal vein embolization (PVE).

DETAILED DESCRIPTION:
ALPPS has been recently proposed as the most effective method to induce marked and rapid hypertrophy of FLR with 95-100% completion rate of the second stage. The most common indication for ALPPS is locally advanced multiple colorectal liver metastases. Unsatisfactory immediate outcomes of ALPPS in surgery of cholangiocarcinoma (CCA) including high mortality reached 48% in patients with h-CCA suggested that patients with biliary cancer should not be treated by ALPPS.

Recently reported modifications of in situ splitting (partial ALPPS, RALPPS (radio-frequency-assisted liver partition with portal vein ligation for staged hepatectomy) and ALTPS (associating liver tourniquet and right portal vein ligation for staged hepatectomy) etc) have been aimed to minimize the operating injury on the first stage, hereby reducing postoperative morbidity.

The other important idea was to preserve all initial benefits of ALPPS in terms of liver hypertrophy and completeness of the second stage. To date, there is no evidence of the benefits of any new ALPPS modification over others in reducing the morbidity of procedure, particularly in patients with CCA..

ELIGIBILITY:
Inclusion Criteria:

* h-CCA, type II-IV, T1-3N0-1M0, volume of FLR<40%
* i-CCA, T1-3N0-1M0, volume of FLR<40%
* Physical status 1-4 according to American Society of Anesthesiologists Physical Status Classification System
* BMI up to 40 kg/m2
* If cirrhosis is present, class A according to Child-Turcotte-Pugh score

Exclusion Criteria:

* h-CCA, stage 4A, B
* i-CCA, stage 4B
* i-CCA, T4N0-1M0
* i-CCA, h-CCA with volume of FLR >45%
* acute cholangitis and/or infected fluid collections, liver abscesses, other unresolved surgical complications of biliary draining procedures.
* jaundice with total bilirubin >50 µmol/L
* prior anamnestic allergic reaction or any other sign of intolerance to iodinated contrast media
* Age under 18 years
* Age above 80 years
* Persons who are incapable of giving consent
* Pregnant or breast-feeding women
* Physical status >4 according to American Society of Anesthesiologists Physical Status Classification System
* BMI > 40 kg/m2
* If cirrhosis is present, class B, C according to Child-Turcotte-Pugh score

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients refered to the Center from other hospitals and primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of Future Liver Remnant (FLR) Hypertrophy | 10 days
  Degree of FLR enlargement (%) with respect to initial volume of FLR [(Post-PVE FLR - Pre-PVE FLR) / (Pre-PVE FLR)] x 100

SECONDARY OUTCOMES:
Major morbidity after the first stage | 10 days
  Grade > II according to Clavien-Dindo classification
Blood loss | intraoperative parameter
  Blood loss during second stage (major liver resection)
Major morbidity after the second stage | 90 days
  Grade > II according to Clavien-Dindo classification
Liver failure | 10 days
  Liver failure after the second stage according to criteria of International Study Group of Liver Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Efanov, Principal Investigator — Moscow Clinical Scientific Center

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03320980/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT03320980/SAP_001.pdf